CLINICAL TRIAL: NCT00969566
Title: Predictive Parameters for Therapeutic Efficacy of Initial Combination Therapy With Sitagliptin and Metformin in Type 2 Diabetic Patients
Brief Title: Predictive Parameters for Efficacy of Sitagliptin and Metformin Combination
Acronym: COSMETIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Soo Lim, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNUBH_ENDO1
Record Dates: First submitted 2009-08-31; First posted 2009-09-01 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: Diabetes
Keywords: Diabetes; Sitagliptin; C-peptide; Glucagon
MeSH Terms: conditions — Diabetes Mellitus | interventions — Sitagliptin Phosphate; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metformin+Sitagliptin (Experimental): Initial combination of metformin and sitagliptin
  Interventions: Drug: sitagliptin, metformin

INTERVENTIONS:
Drug: sitagliptin, metformin — sitagliptin 100mg once daily and metformin 500mg twice daily, orally, for 24 weeks.
  Other Names: Januvia

SUMMARY:
It is well established that inhibition of dipeptidyl peptidase (DPP)-IV reduces glucose levels in both fasting and postprandial states and preserves pancreatic beta cell function in patients with type 2 diabetes. Their mechanism of action is derived from increased incretin (GLP-1) levels, which stimulate insulin secretion as well as insulin biosynthesis and inhibit glucagon secretion from pancreas. Recent studies reported that combination therapy with DPP-IV inhibitors and metformin have additive or synergistic effects in lowering glycose level, preserving beta-cell mass and function as well as enhancing insulin sensitivity. However, there have been few studies about the difference of glucose lowering effect of combination therapy of DPP-IV inhibitors and metformin according to the secretory capacity of pancreas.

The researchers hypothesized that combination therapy with DPP-IV inhibitor and metformin may have more favorable glucose lowering effect in type 2 diabetic patients who have preserved pancreatic secretory function. The researchers plan to investigate the difference of glucose lowering effect of 24 weeks treatment with sitagliptin (DPP-IV inhibitor) in combination with metformin according to basal c-peptide and glucagon level in type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* HbA1c ≥ 7%
* Age ≥ 18

Exclusion Criteria:

* Contraindication to sitagliptin or metformin
* Pregnant or breast feeding women
* Reproductive-age women who refuse contraception
* Type 1 diabetes, gestational diabetes, or diabetes with secondary cause
* Chronic hepatitis B or C (except healthy carrier of HBV), liver disease (AST/ALT > 3-fold the upper limit of normal)
* Renal failure (Cr > 2.0)
* Cancer within 5 years (except squamous cell cancer, cervical cancer, thyroid cancer with appropriate treatment)
* Not appropriate for oral antidiabetic agent
* Medication which affect glycemic control
* Disease which affect efficacy and safety of drugs
* Other clinical trial within 30 days

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-01; Primary Completion 2010-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
The change of HbA1c | 52 weeks

SECONDARY OUTCOMES:
Fasting Plasma Glucose (FPG) | 52 weeks
Postprandial Plasma Glucose (PPG) | 52 weeks
C-peptide | 52 weeks
Glucagon | 52 weeks
Homeostatic model assessment of insulin resistance (HOMA-IR) | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Soo Lim, MD, MPH, PHD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea